CLINICAL TRIAL: NCT06786754
Title: FIBROBLASTS AND THORACIC AORTIC ANEURYSMS: IN VITRO CHARACTERIZATION IN PATIENTS WITH MARFAN SYNDROME AND GENETIC AORTIC DISEASES
Brief Title: Fibroblasts and Thoracic Aortic Aneurysms: in Vitro Characterization in With Marfan Syndrome and Genetic Aortic Diseases
Acronym: FIBRA
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: FIBRA
Record Dates: First submitted 2025-01-09; First posted 2025-01-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Rare Diseases; Thoracic Aortic Aneurysm (TAA); Marfan Syndrome
Keywords: Fibroblasts; Collagen turnover; thoracic aortic aneuryms
MeSH Terms: conditions — Rare Diseases; Aortic Aneurysm, Thoracic; Marfan Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Fibroblasts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Syndromic TAA: Presence of thoracic aortic aneurysms and pleiotropic effects
- Non-syndromic TAA: Presence of thoracic aortic aneurysms without pleiotropic effects
- Healthy Controls: healthy volunteers from the general population, matched fro age with the two case groups

SUMMARY:
The aim of the present study is to characterise the phenotype of fibroblasts and to classify different mechanisms involved in the onset and progression of TAAD in syndromic and non-syndromic subjects in order to evaluate potential markers related to TAAD.

DETAILED DESCRIPTION:
The aim of the study is to analyse cutaneous fibroblast properties in patients with thoracic aortic aneurysms (both syndromic and non-syndromic) to identify differences in molecular mechanisms in collagen turnover pathways compared to healthy controls in the general population.

ELIGIBILITY:
Inclusion Criteria (general for the study):

signed informed consent; subjects aged 18 years and above.

Inclusion Criteria (Case):

subjects with Marfan syndrome and thoracic aortic aneurysms (in clinical follow-up or with cardiac surgery program); subjects with non-syndromic thoracic aortic aneurysms (in clinical follow-up or with cardiac surgery program);

Inclusion Criteria (healthy controls):

absence of any aortic/thoracic disease;

Exclusion Criteria (all groups):

* Presence of any confounding cardiovascular risk factor (hypertension, dyslipidaemia, diabetes, smoking habits) or previous cardiovascular disease
* Corticosteroid or Steroids or Fluorochinolones treatment within six months before enrollment Subjects on chronic immunosuppressive therapies such as oral steroids, but also on chronic topical steroids in the area of investigation;
* A history of keloid formation (data found in anamnesis and medical records);
* Anaesthetic drug allergy (data found in anamnesis and medical records).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: resaerch hospital for rare cardiovascular diseases
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Fibroblasts phenotype: cell morphology and migration | 12 months
  cell morphology: phase-contrast microscopy
Fibroblasts phenotype: cell morphology and migration | 12 months
  Cell migration: wound healing assay (scratch test).

SECONDARY OUTCOMES:
Expression of genes and proteins involved in collagen turnover and extracellular matrix remodeling pathways | 16 months
  mRNA extraction and real-time PCR to assess the expression of genes involved in collagen turnover;
Expression of genes and proteins involved in collagen turnover and extracellular matrix remodeling pathways | 16 months
  Slot blot to assess ECM proteins and degrading proteases.
Levels of metalloproteinases involved in ECM degradation | 24 months
  SDS-zymography

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Genetic Centre IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
IPD sharing will be defined at the active enrolment process of the study

REFERENCES:
- [Background] Ignotz RA, Massague J. Transforming growth factor-beta stimulates the expression of fibronectin and collagen and their incorporation into the extracellular matrix. J Biol Chem. 1986 Mar 25;261(9):4337-45. PMID 3456347
- [Background] Lu P, Takai K, Weaver VM, Werb Z. Extracellular matrix degradation and remodeling in development and disease. Cold Spring Harb Perspect Biol. 2011 Dec 1;3(12):a005058. doi: 10.1101/cshperspect.a005058. PMID 21917992
- [Background] Plikus MV, Wang X, Sinha S, Forte E, Thompson SM, Herzog EL, Driskell RR, Rosenthal N, Biernaskie J, Horsley V. Fibroblasts: Origins, definitions, and functions in health and disease. Cell. 2021 Jul 22;184(15):3852-3872. doi: 10.1016/j.cell.2021.06.024. PMID 34297930